CLINICAL TRIAL: NCT00734695
Title: The Effect of Subconjunctival Vitamin c on Recovery Rate and End Result From Eye Burn.
Brief Title: Comparing the Use of Vitamin c (Ascorbic Acid) in Eye Burn in Subconjunctival Injection to Topical or Oral Treatment.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: couldn't recruit patients
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Collaborators: Rambam Health Care Campus (Other); Soroka University Medical Center (Other)
Responsible Party: Modi Naftali, Baruch Pade Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: vitcbrn.CTIL
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Burn
Keywords: BURN; EYE; VITAMIN C; ASCORBIC ACID
MeSH Terms: conditions — Burns | interventions — Ascorbic Acid; Vision, Ocular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Baruch Pade Medical Center
  Interventions: Dietary Supplement: vitamin c
- 2 (Active Comparator): Rambam Medical Center
  Interventions: Dietary Supplement: vitamin c
- 3 (Active Comparator): Soroka Medical Center
  Interventions: Dietary Supplement: vitamin c

INTERVENTIONS:
Dietary Supplement: vitamin c — Subconjunctival daily or bid
  Other Names: subconjunctival; ascorbic acid
  Arms: 1
Dietary Supplement: vitamin c — topical and systemic
  Other Names: Burn; eye; ascorbic acid
  Arms: 2
Dietary Supplement: vitamin c — topical systemic
  Other Names: burn
  Arms: 3

SUMMARY:
Eye burns may cause a severe permanent damage. One kind of treatment is the use of vitamin C (Ascorbic acid). This study will compare between subconjunctival topical and/or systemic route of administration and topical and/or systemic administration.

DETAILED DESCRIPTION:
In order to prevent permanent and severe damage to the eye after eye burn early treatment is mandatory. It is well known and published that the use of Vitamin c may contribute to the healing process of such burns, including burns from chemicals or heat. We believe that the route pf administration of the medicine is as important as the kind of medicine and that subconjunctival injection will have better effect and will influence in a favorable manner on the the end result as well as on the time of the healing.

In order to be able to compare between cases we made a new definition of the severity of the burn according to the extension of the damage on the cornea, conjunctiva and limbus, and according to the severity and depth of the ischemia.

In 3 medical centers 3 protocols of treatment and followup will be compared while only in Baruch Pade Medical Center the main route of administration will be subconjunctival on top of the topical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Eyes clinic patients presented with acute chemical or thermal burn.

Exclusion Criteria:other disease

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-11 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
EXTENSION OF FLORSCEIN PAINT ON THE CORNEA AND CONJUNCTIVA | BID

CONTACTS AND LOCATIONS:
Overall Officials: naftali modi, MD, Principal Investigator — Baruch Pade medical center
Locations (2):
- Israel (2):
  - Movshovitz Ina, Afula
  - Naftali Modi, Tiberias